CLINICAL TRIAL: NCT07139977
Title: Open-Label Phase II Trial of Enfortumab Vedotin in Recurrent or Persistent Endometrial Carcinoma
Brief Title: Study of EV for Recurrent Endometrial Carcinoma
Acronym: EV-4-EC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: William Bradley (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor-Investigator, William Bradley, Professor, Obstetrics and Gynecology, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00055484
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; endometrioid; serous endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enfortumab vedotin: 1.25 mg/kg on days 1,8, and 15 of the 28 day cycle (Experimental): Single arm trial
  Interventions: Drug: Enfortumab Vedotin

INTERVENTIONS:
Drug: Enfortumab Vedotin — Enfortumab vedotin is an ADC comprised of a fully human IgG1Κ antibody conjugated to the microtubule-disrupting agent MMAE via a protease-cleavable linker. Enfortumab vedotin is thought to induce anti-tumor activity by binding to the nectin-4 protein on the surface of cancer cells, leading to internalization, proteolytic cleavage of the linker, and intracellular release of MMAE that subsequently disrupts tubulin polymerization and leads to mitotic arrest and apoptosis of the tumor cell.

SUMMARY:
This study is testing a drug called enfortumab vedotin in up to 12 patients with advanced endometrial (uterine) cancer that has worsened after previous treatments, including immunotherapy. The goal is to see how well the drug works and how safe it is. Patients will be treated for up to one year and followed over time to monitor their health and response to the treatment.

DETAILED DESCRIPTION:
This is an open-label, single-arm Phase II trial evaluating the efficacy and safety of enfortumab vedotin monotherapy in up to 12 patients with advanced or metastatic endometrial carcinoma who have progressed after prior chemotherapy and anti-PD-1 or other immunotherapy. Treatment will continue for up to 12 months or until disease progression per RECIST v1.1, unacceptable toxicity, or patient withdrawal.

Patients with stable disease or objective response may remain on therapy unless discontinued due to toxicity or patient choice. Those who discontinue treatment for reasons other than progression will be followed for disease status until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient of age ≥18 years.
2. Recurrent and progressive endometrial cancer, all stages at primary diagnosis. The histology types will be pending the preclinical assessments, but can include:

   1. Endometrioid endometrial carcinoma
   2. Serous endometrial carcinoma
3. Prior standard of care of surgical intervention, including hysterectomy.
4. Evidence of disease progression on or following the most recent line of therapy prior to screening. Therapy must include platinum-based chemotherapy. If the patient is eligible for immunotherapy, this must have been provided. Patient may have received either radiation therapy or hormone therapy, neither of which will be considered a line of therapy. Chemotherapy during radiotherapy will not be considered a line of therapy.
5. Maximum of three prior lines of therapy. Neo-adjuvant and postsurgical therapy, if provided, will be counted as 1 line of therapy. Therapy given in a maintenance fashion after primary treatment will not be counted as a line of therapy.
6. IHC expression of nectin-4.
7. Toxicity from prior treatment recovered to G1 or G0.
8. ECOG status of 1 or 0.
9. At least 1 measurable target lesion according to RECIST v1.1, including the following criteria:

   1. Non-nodal lesion that measures ≥ 1.0 cm in the longest diameter.
   2. Lymph node (LN) lesion that measures as ≥ 1.5 cm in the short axis.
   3. The lesion is suitable for repeat measurement using computed tomography/magnetic resonance imaging (CT/MRI). Lesions that have had external beam radiotherapy (EBRT) or locoregional therapy must show radiographic evidence of subsequent growth after treatment.
10. Documented tumor status for MSI and MMR.
11. In the opinion of the investigator, the patient must have a life expectancy of at least 12 weeks and be well enough to receive experimental therapy.
12. Adequate organ function as determined by laboratory tests defined in the table below at screening.

    Hematological: Absolutely neutrophil count (ANC)≥ 1500/μL, Platelets ≥ 100,000/μL, Hemoglobin ≥ 9.0 g/dL or 5.6 mmol/L, No erythropoietin dependency or packed red blood cell transfusion within last 2 weeks.

    Renal: Creatinine, OR ≤ 1.5 x ULN, Creatinine clearance as calculated per institutional standard ≥ 30 mL/min for patients with creatinine > 1.5 × institutional ULN Hepatic: Total bilirubin ≤ 1.5 × upper limit of normal (ULN) ≤ 3 ULN for participants with Gilbert's syndrome. AST, ALT ≤ 3 × ULN (≤ 5 × ULN for participants with liver metastases
13. Ability to understand a written informed consent document, and the willingness to sign it.
14. Pregnancy: It is not known what effects this treatment has on human pregnancy or development of the embryo or fetus. Therefore, female patients participating in this study should avoid becoming pregnant, and male patients should avoid impregnating a female partner. Nonsterilized female patients of reproductive age and male patients should use effective methods of contraception through defined periods during and after study treatment as specified below. Female patients must meet one of the following:

    1. Postmenopausal for at least one year before the screening visit, or
    2. Surgically sterile, or
    3. If they are of childbearing potential, agree to practice two effective methods of contraception from the time of signing of the informed consent form through three months after the last dose of study drug, AND
    4. Must also adhere to the guidelines of any treatment specific pregnancy prevention program, if applicable, or
    5. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.) Male patients/partners of patients, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the following:

    <!-- -->

    1. Practice effective barrier contraception during the entire study treatment period and through 90 days after the last study drug dose, OR
    2. Must also adhere to the guidelines of any treatment specific pregnancy prevention program, if applicable, OR
    3. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

1. Diagnosis of endometrial sarcoma (leiomyosarcoma, endometrial stromal sarcoma, high-grade sarcoma).
2. Diagnosis of non-endometrioid and non-serous endometrial cancer. Mixed tumors involving histologic types other than serous and endometrioid will not be eligible.
3. Tumor sample does not express nectin-4 (local IHC testing).
4. Symptomatic CNS metastases or leptomeningeal metastases. Patients with symptomatic brain metastasis must be treated and must be stable for at least 4 weeks prior to study treatment.
5. Active second malignancy with anti-cancer treatments (except for treated in-situ carcinomas [e.g., breast, cervix, bladder], or basal or squamous cell carcinoma of the skin) within the past 24 months.
6. Sensory or motor neuropathy ≥ G2
7. Prior history of significant cardiovascular impairment within 12 months of the first dose of study drug: such as history of congestive heart failure greater than New York Heart Association (NYHA)Class II, unstable angina, myocardial infarction, or cerebrovascular accident (CVA) stroke, or cardiac arrhythmia associated with hemodynamic instability.
8. Active infection requiring systemic IV antibiotics within 14 days, or oral antibiotics within 7 days, prior to administration of study drugs. Regular treatment of urinary tract infection (UTI) and/or topical treatment are allowed.
9. Uncontrolled diabetes defined as HgbA1c of ≥ 8%.
10. Hepatitis B, C, or HIV infection.
11. Have not recovered to CTCAE v5.0 Grade 0 or 1 (except chemotherapy related grade 2 peripheral neuropathy, or grade 2 endocrinopathy with adequate replacement therapy) from any toxicity and/or complications from major surgery or prior cancer therapeutics before starting therapy.
12. Ongoing treatment for EC, including radiation therapy, hormonal therapy, chemotherapy, immunotherapy, or any investigational therapy, unless they have been discontinued at least 4 weeks prior to screening and there is no plan to re-initiate during the study. radiation therapy is allowed prior to and during study drug administration as long as there are no acute toxicities.
13. Active intestinal obstruction.
14. Known psychiatric or substance use disorders that would interfere with cooperation with the requirements of the trial.
15. Any conditions that required systemic immunosuppression therapy (in dosing exceeding 10 mg daily of prednisone or equivalent) within 7 days prior to the first dose of study drug.
16. Pregnant or lactating patients.
17. In the opinion of the Investigator, have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study or make study participation, not in the best interest of the patient. The Investigator should discuss with the Sponsor and/or study leaders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Estimate the overall response rate (ORR) | 24 months
  Overall response rate (ORR) of enfortumab vedotin treatment for patients with endometrioid or serous endometrial cancer, i.e., proportion of patients with a complete or partial response as per RECIST v1.1.
Evaluate the safety of enfortumab vedotin treatment | 24 months
  Incidence of adverse events (AEs) and serious adverse event (SAEs) as defined by NCI CTCAE v5.

SECONDARY OUTCOMES:
Characterize the Duration of Response (DOR) | 30 months
  Duration of response (DOR), i.e., the time from date of initial response to therapy by RECIST v1.1 to subsequent disease progression, relapse or death.
Estimate overall survival (OS) | 24 months
  Median overall survival (OS), i.e., the time from date of treatment to the date of death due to any reason.
Estimate progression-free survival (PFS) | 12 months
  the time from date of treatment to the date of disease progression or death, as assessed per RECIST v1.1.
Duration of response (DOR) by MMR status. | 30 months
  Subgroup analysis of response by MMR status (i.e., proficient or deficient), and by TCGA sub-type, 1. Ultramutated (POLE), 2. Hypermutated (MSI), 3. Copy Number low (endometrioid), 4. Copy-Number high (serous like).

CONTACTS AND LOCATIONS:
Overall Officials: William Bradley, MD, Principal Investigator — Medical College of Wiscnson
Locations (1):
- Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
This is a single-site, Investigator-Initiated Trial (IIT). There are no plans to share individual participant data beyond the study site.